CLINICAL TRIAL: NCT07374549
Title: A Randomized, Open-Label, Controlled, Multicenter Phase 2 Trial of SYS6002 Versus PADCEV in Patients With Advanced Urothelial Carcinoma
Brief Title: SYS6002 vs PADCEV in Patients With Advanced Urothelial Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CSPC Megalith Biopharmaceutical Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYS6002-00X
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Advanced Urothelial Carcinoma
MeSH Terms: interventions — enfortumab vedotin

STUDY DESIGN:
Intervention Model Description: Participants in this trial will be randomly assigned to one of two groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SYS6002 (Active Comparator)
  Interventions: Drug: SYS6002
- enfortumab vedotin (Active Comparator): enfortumab vedotin monotherapy
  Interventions: Drug: enfortumab vedotin

INTERVENTIONS:
Drug: SYS6002 — SYS6002 by intravenous (IV)
  Arms: SYS6002
Drug: enfortumab vedotin — 1.25 mg/kg by IV on Day 1、8、15, every 28 days.
  Arms: enfortumab vedotin

SUMMARY:
This study is a randomized, open-label, controlled, multicenter phase II clinical trial, which aims to evaluate the safety and efficacy of SYS6002 versus enfortumab vedotin in the treatment of participants with advanced urothelial carcinoma.

This study has not yet been submitted for ethical review. The current registration is a pre-registration. Recruitment will be initiated only after formal approval is obtained from the relevant Ethics Committee or Institutional Review Board.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients aged 18-80 years (inclusive);
* 2. Pathologically confirmed patients with advanced urothelial carcinoma who have received a platinum-based chemotherapy with anti-PD-(L)1 agent. For those who received these therapies in the adjuvant or neoadjuvant setting, disease progression must have occurred during treatment or within 12 months of treatment completion;
* 3 An archival tumor tissue sample or a fresh tissue sample should be provided;
* 4 Subjects must have measurable disease according to RECIST (version 1.1);
* 5 Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* 6 Life expectancy of ≥ 3 months;
* 7 Major organ function must meet the relevant laboratory test standards for hematology, renal function, liver function, and coagulation within 7 days prior to treatment;
* 8Sexually active fertile subjects must agree to use methods of contraception during the study and at least 7 months after termination of study therapy and have a negative urine or serum pregnancy test within 7 days prior to randomization;
* 9.Willing to participate in the study, understand the study procedures, and sign a written informed consent form.

Exclusion Criteria:

* 1.Active central nervous system metastases or leptomeningeal metastasis;
* 2.Adverse events from prior anti-tumor therapy not recovered to ≤ Grade 1 (unless the investigator deems there is no safety risk)；
* 3.Any serious and/or uncontrolled concurrent illness that may interfere with patient's participation in the study:

  1. Participants with a history of severe cardiovascular disease within 6 months prior to randomization, including but not limited to:

     Severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia and third-degree atrioventricular block requiring clinical intervention; corrected QT interval > 480 ms by Fridericia method (Fridericia formula: QTcF = QT/RR^0.33, RR = 60/heart rate); With history of myocardial infarction, unstable angina pectoris, angioplasty and coronary artery bypass surgery; New York Heart Association (NYHA) classification Grade III and above heart failure, and left ventricular ejection fraction (LVEF) < 50% in the tests and examinations during the screening period; cerebrovascular accidents; pulmonary embolisms;
  2. Other clinically significant diseases:

HbA1c > 8%; Participants with active keratitis and corneal ulcer, or fundus lesions with a risk of blindness; Grade ≥2 neuropathy prior to randomization; Severe infection within 4 weeks prior to randomization; active infection requiring systemic antibiotics, antiviral, or antifungal therapy within 2 weeks prior to randomization; Active HBV or HCV infection; History of immunodeficiency (HIV-positive, acquired or congenital immunodeficiency, etc.), or organ transplantation; History of another malignancy within 3 years prior to randomization; History of interstitial lung disease (ILD) / non-infectious pneumonia, or current ILD/non-infectious pneumonia, or imaging findings at screening that cannot rule out these conditions, except for those who are determined to be risk-free after discussion between the investigator and the sponsor; Pleural effusion, ascites or pericardial effusion with symptoms or requiring puncture or drainage within 2 weeks prior to randomization;

* 4.Use of other unmarketed clinical investigational drugs or treatments, chemotherapy, radiotherapy targeted therapy within 4 weeks prior to randomization; use of traditional Chinese medicine with anticancer indication, oral fluoropyrimidine drugs, small molecule targeted drug within 2 weeks prior to randomization; use of palliative radiation or local therapy within 2 weeks prior to randomization;with major surgery within 4 weeks prior to randomization;
* 5.Allergy to any component of SYS6002, or humanized monoclonal antibodies; investigator-determined ineligibility for enfortumab vedotin therapy.
* 6. Other conditions deemed by the investigator as unsuitable for participation in this clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-06-20 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence and frequency of Adverse Event (AE) | Up to approximately 2 years

SECONDARY OUTCOMES:
Incidence of treatment-related peripheral neuropathy and≥1-grade worsening in treatment-related peripheral neuropathy from baseline | Up to 2 years
Incidence of treatment-related hyperglycemia | Up to 2 years
Incidence of treatment-related cutaneous adverse reactions | Up to 2 years
Objective Response Rate (ORR) | Up to 2 years
  Objective response rate is defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) per RECIST v.1.1.
Duration of Response (DOR) | Up to 2 years
  DOR is defined as the time from the date of the first confirmed objective response (CR or PR that is subsequently confirmed) to the date of the first documented disease progression (PD) per RECIST v1.1 or death from any cause, whichever occurs first
Disease Control Rate (DCR) | :Up to 2 years
  The percentage of participants who experience a best response of CR, PR or stable disease (SD).
Progression Free Survival (PFS) | Up to 2 years
  PFS is defined as the time from the date of randomization to the first documentation of PD as assessed by investigator per RECIST v.1.1, or death due to any cause, whichever occurs earlier.
Overall Survival | Up to 2 years